CLINICAL TRIAL: NCT05318391
Title: Translational Study of Molecular Classification of Relapsed/Refractory Diffuse Large B-cell Lymphoma
Status: Completed | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Wuxi People's Hospital (Other); Shanghai Minhang Central Hospital (Other)
Responsible Party: Principal Investigator, Peng Liu, Chief of hematology department, Shanghai Zhongshan Hospital
Other Study IDs: SHZS-DLBCL001
Record Dates: First submitted 2021-05-08; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Lymphoma, Large B-Cell, Diffuse; Gene Expression Profiling
Keywords: Canhelp-COO Assay
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Transcriptome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Formalin-Fixed and Parrffin-Embedded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group/Cohort: Retrospective Cohort： Participants who diagnosed with relapsed/refractory diffuse large B-cell lymphoma (R/R DLBCL) patients and treated with BTK inhibitor or lenalidomide and its biosimilars.
  Interventions: Diagnostic Test: Gene expression profile

INTERVENTIONS:
Diagnostic Test: Gene expression profile — Diagnostic Test:
  The Canhelp-COO Assay (Canhelp Genomics CO., Ltd) for differentiating COO subtypes using gene expression analysis by real-time PCR (RT-PCR)

SUMMARY:
The purpose of the study is to investigate the proportion of the cell-of-origin (COO) subtypes in relapsed/refractory diffuse large B-cell lymphoma (R/R DLBCL) treated with BTK inhibitor or lenalidomide and its biosimilars.

DETAILED DESCRIPTION:
This is a multi-center, observational, retrospective study that examines approximately 200 R/R DLBCL patients treated with BTK inhibitors or lenalidomide and its biosimilars. For patients meet the inclusion criteria, gene expression analysis is performed on formalin fixed paraffin-embedded tissue by using Canhelp-COO Assay, and determine the COO subtype for each specimen. The proportion of COO subtypes in R/R DLBCL and the correlation between COO subtypes and clinicopathological information are further analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed diagnosis of DLBCL, including transformed large B-cell lymphoma from previous indolent lymphoma.
2. Meet the definition of relapsed/refractory DLBCL.
3. Patients received BTK inhibitors and/or lenalidomide and its biosimilars after the failure of the first-line standard treatment. The efficacy was evaluated by the investigators. Cohort plans to enroll one hundred patients with BTK inhibitors treatment (excluding the combination with lenalidomide), one hundred patients with lenalidomide treatment (excluding the combination with BTK inhibitors) and any number of the cases with BTK inhibitors and lenalidomide combination.

   a) BTK inhibitors include ibrutinib, zanubrutinib and acalabrutinib
4. Patients with comprehensive history information and follow-up data.
5. Patient able to provide written informed consent, agreeing that the donated samples and related information can be used for all medical research.

Exclusion Criteria:

1. The archived tumor tissue is too little to test.
2. Patients with primary central nerve system large B-cell lymphoma or primary mediastinal large B-cell lymphoma.
3. R/R DLBCL patients receive BTK inhibitor or lenalidomide treatment for less than one cycle.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Relapsed/refractory DLBCL patients who had received BTK inhibitors and/or lenalidomide and its biosimilars after the failure of the first-line standard treatment.Patients with comprehensive history information and follow-up data and are able to provide written informed consent, agreeing that the donated samples and related information can be used for all medical research.
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
proportion of the cell of origin subtypes in the study population | up to 24 weeks
  Investigate the proportion of the cell of origin (COO) subtypes in relapsed/refractory diffuse large B-cell lymphoma (R/R DLBCL) treated with BTK inhibitor or lenalidomide and its biosimilars.

SECONDARY OUTCOMES:
correlation between COO subtypes and the ORR of the treatment of R/R DLBCL. | up to 24 weeks
  Based on the objective response rate (ORR) measured by the investigator, explore the correlation between COO subtypes and the efficacy of BTK inhibitors, lenalidomide and its biosimilars in the treatment of R/R DLBCL.
correlation between COO subtypes and the PFS and OS of the treatment of R/R DLBCL. | up to 24 weeks
  Based on the progression-free survival (PFS) and overall survival (OS) measuredd by the investigator, explore the correlation between COO subtypes and the efficacy of BTK inhibitors, lenalidomide and its biosimilars in the treatment of R/R DLBCL .

CONTACTS AND LOCATIONS:
Overall Officials: Peng Liu, MD,PhD, Principal Investigator — Fudan University
Locations (1):
- Yian Zhang, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yan WH, Jiang XN, Wang WG, Sun YF, Wo YX, Luo ZZ, Xu QH, Zhou XY, Cao JN, Hong XN, Li XQ. Cell-of-Origin Subtyping of Diffuse Large B-Cell Lymphoma by Using a qPCR-based Gene Expression Assay on Formalin-Fixed Paraffin-Embedded Tissues. Front Oncol. 2020 Jun 5;10:803. doi: 10.3389/fonc.2020.00803. eCollection 2020. PMID 32582543